CLINICAL TRIAL: NCT01457807
Title: A Phase I, Single-centre, Double-blind, Randomised, Placebo-controlled, Parallel Group Study to Assess the Pharmacokinetics, Safety and Tolerability of Two Different Extended Release Formulations of Tablets of AZD3241 (300 mg) After Administration of Multiple Doses in Healthy Male and Female Volunteers
Brief Title: To Assess the Effect of Administration of 2 Formulation of AZD3241 on Blood Concentration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: D0490C00003
Record Dates: First submitted 2011-10-10; First posted 2011-10-24 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Parkinson's Disease
Keywords: Phase 1; Parkinson's disease; pharmacodynamic; biomarkers; pharmacokinetics; extended release formulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): AZD3241 300mg extended release formulation 1
  Interventions: Drug: AZD3241 ER formulation 1; Drug: AZD3241 Alternative titration scheme with formulation 1 or 2
- 2 (Experimental): AZD3241 300mg extended release formulation 2
  Interventions: Drug: AZD3241 Alternative titration scheme with formulation 1 or 2
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3241 ER formulation 1 — Oral tablets, 100mg bd on Day 1 to Day 2, 200mg bd on Day3, 300mg bd on Day 4 to Day7 and 300mg Once daily on Day 8 with High Fat Breakfast
  Arms: 1
Drug: Placebo — Placebo will be administered with the same intervention scheme as intervention 1 and 2
  Arms: 3
Drug: AZD3241 Alternative titration scheme with formulation 1 or 2 — 50 mg oral dose bd on Day 1, 100 mg oral dose bd on Day 2 and 3, 200 mg oral dose bd on Day 4, 300 mg oral dose bd on Day 5 to 7 and 300 mg once in the morning on Day 8
  Other Names: This titration scheme will only be used if ER formulations 1 or 2 are not well tolerated
  Arms: 1; 2

SUMMARY:
To evaluate the pharmacokinetics of AZD3241 following multiple administration of 2 new, different extended release formulations of tablets of AZD3241 (300 mg), in relation to the 100 mg extended release tablet used in a previous study and potential food interaction. The safety and tolerability of AZD 3241 will also be investigated as a secondary objective. In addition to these a number of exploratory objectives will be investigated with blood sampling.

DETAILED DESCRIPTION:
A Phase I, Single-centre, Double-blind, Randomised, Placebo-controlled, Parallel Group Study to Assess the Pharmacokinetics, Safety and Tolerability of Two Different Extended Release Formulations of Tablets of AZD3241 (300 mg) after Administration of Multiple Doses in Healthy Male and Female Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male or female volunteers aged 30 to 65 years, inclusive, with suitable veins for cannulation or repeated venepuncture
* Female volunteers must have a negative pregnancy test at Screening and on admission to the CPU, must not be lactating and must be of non childbearing potential, confirmed at Screening
* Male volunteers must be willing to use barrier contraception ie, condoms, from the first day of dose administration until 3 months after the last dose of the IP
* Volunteers must have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD3241
* Orthostatic hypotension defined as 25 mmHg decrease in systolic and/or 15 mmHg decrease in diastolic BP as measured at enrolment and/or randomisation
* History of intolerance or hypersensitivity to mannitol
* Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF)>450 ms or shortened QTcF<340 ms or a family history of long QT syndrome
* Abnormal vital signs, after 10 minutes of rest in supine position, defined as any of the following:Systolic BP>140 mmHg., Diastolic BP>90 mmHg., Heart rate<40 or >85 beats per minute.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
AUC(0-12),ss: Area under the plasma concentration-time curve from time zero to the end of the 12-hour dosing interval at steady state. | Day 1 until 24 hours post last dose (administered on the morning of Day 8)
AUC(0-12),ss/DN: Area under the plasma concentration-time curve from time zero to the end of the 12-hour dosing interval at steady state observed with the 300 mg ER formulations normalised to a 100 mg dose of AZD3241 | Day 1 until 24 hours post last dose (administered on the morning of Day 8)
Css,max: Observed maximum plasma concentration at steady state.Css,max/DN Observed maximum plasma concentration at steady state observed with the 300 mg ER formulations normalised to a 100 mg dose of AZD3241. | Day 1 until 24 hours post last dose (administered on the morning of Day 8)
Css,min: Observed minimum plasma concentration at steady state.Css,min/DN Observed minimum plasma concentration at steady state observed with the 300 mg ER formulations normalised to a 100 mg dose of AZD3241. | Day 1 until 24 hours post last dose (administered on the morning of Day 8)
Css,av: Average plasma concentration during the 12-hour dosing interval at steady state calculated as follows: AUC(0-12),ss/12 h. | Day 1 until 24 hours post last dose (administered on the morning of Day 8)
Description of fluctuation at steady-state [(Css,max-Css,min)/Css,av] | Day 1 until 24 hours post last dose (administered on the morning of Day 8)
AUC(0-t),ss: Area under the plasma concentration-time curve from time zero to the last quantifiable time point. | Day 1 until 24 hours post last dose (administered on the morning of Day 8)
λz,ss: Terminal elimination rate constant at steady state. | Day 1 until 24 hours post last dose (administered on the morning of Day 8)
t½λz,ss: Half-life of terminal elimination phase at steady state. | Day 1 until 24 hours post last dose (administered on the morning of Day 8)

SECONDARY OUTCOMES:
Description of the safety and tolerability profile in terms of Adverse Events of 8 days of administration of AZD3241, up to steady state (300 mg twice daily), of 2 new, different extended release tablets of AZD3241 (300 mg), including initial titration. | Day 1 to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Quintiles drug research unit, 6 Newcomen Street, SE1 1YR; Bjorn Paulsson, MD, PHD, Study Director — Astra Zeneca, Sodertalje, Sweden; Bo Fransson, MD, PHD, Study Chair — Astra Zeneca, Sodertalje, Sweden
Locations (1):
- Research site, London, United Kingdom